CLINICAL TRIAL: NCT00412568
Title: Evaluation of Conventional Photorefractive Keratectomy (PRK) in U.S. Army Personnel, Substudy of: Initial Evaluation of Excimer Laser Keratorefractive Surgery in U.S. Army Personnel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Collaborators: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WRAMC WU # 04-2335-99d; WU #2335-99 (master protocol)
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2007-11

CONDITIONS: Myopia
Keywords: Naturally occuring myopia with or without astigmatism.
MeSH Terms: conditions — Myopia | interventions — Photorefractive Keratectomy

ARMS (1):
- 1 (Active Comparator): PRK control group
  Interventions: Procedure: Photorefractive Keratectomy (PRK)

INTERVENTIONS:
Procedure: Photorefractive Keratectomy (PRK) — vision correction with PRK

SUMMARY:
The purpose of this study is to:

1. evaluate the safety and efficacy of conventional PRK in U.S. Army personnel who have naturally occurring myopia with or without astigmatism.
2. compare the data from this control group to study groups undergoing wavefront guided PRK.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, of any race, and at least 21 years old at the time of the pre-operative examination, and have signed an informed consent. The lower age limit of 21 years is intended to ensure documentation of refractive stability.
2. Manifest refractive spherical equivalent (MSE) of up to 6.00 diopters (D) at the spectacle plane with refractive cylinder up to 3.00 D.
3. Manifest refraction and LADARWave™ refractions must be within 1.00 D.
4. Best spectacle corrected visual acuity of 20/20 or better in both eyes.
5. Demonstrated refractive stability, confirmed by clinical records. Neither the spherical nor the cylindrical portion of the refraction may have changed more than 0.50D during the 12-month period immediately preceding the baseline examination, as confirmed by clinical records.
6. Soft contact lens users must have removed their lenses at least 2 weeks before baseline measurements. Hard contact lens users (PMMA or rigid gas permeable lenses) must have removed their lenses at least 4 weeks prior to baseline measurements and have 2 central keratometry readings and 2 manifest refractions taken at least 1 week apart that do not differ by more than 0.50 D in either meridian; mires should be regular.
7. Located in the greater Washington DC area for a 12-month period.
8. Consent of the subject's command (active duty) to participate in the study.
9. Access to transportation to meet follow-up requirements.

Exclusion Criteria:

1. Female subjects who are pregnant, breast-feeding or intend to become pregnant during the study. Female subjects will be given a urine pregnancy test prior to participating in the study to rule out pregnancy.
2. Concurrent topical or systemic medications that may impair healing, including corticosteroids, antimetabolites, isotretinoin (Accutane), amiodarone hydrochloride (Cordarone) and/or sumatripin (Imitrex).
3. Medical condition(s), which, in the judgment of the investigator, may impair healing, including but not limited to: collagen vascular disease, autoimmune disease, immunodeficiency diseases, and ocular herpes zoster or simplex.
4. Active ophthalmic disease, neovascularization of the cornea within 1mm of the intended ablation zone, or clinically significant lens opacity.
5. Evidence of glaucoma or an intraocular pressure greater than 22 mm Hg at baseline.
6. Evidence of keratoconus, corneal irregularity, or abnormal videokeratography in either eye.
7. History of recurrent erosions or epithelial basement dystrophy.
8. Patients with known sensitivity or inappropriate responsiveness to any of the medications used in the post-operative course.
9. Any physical or mental impairment that would preclude participation in any of the examinations.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2004-05; Study Completion 2008-03

PRIMARY OUTCOMES:
safety, efficacy, and refractive stability | one year after procedure

CONTACTS AND LOCATIONS:
Overall Officials: KRAIG S. BOWER, MD, Principal Investigator — Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Center For Refractive Surgery, Washington D.C., District of Columbia, United States